CLINICAL TRIAL: NCT04837586
Title: Self-weighing for Weight Management in Adolescents Seeking Obesity Treatment: A Randomized Pilot
Brief Title: Self-Weighing for Adolescents Seeking Obesity Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2021-29697
Record Dates: First submitted 2021-03-30; First posted 2021-04-08 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Adolescent Obesity
Keywords: Obesity
MeSH Terms: conditions — Pediatric Obesity; Obesity | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard Care (Active Comparator): Individuals in this arm will receive standard care for their obesity in the Pediatric Weight Management Clinic
  Interventions: Other: Standard Care
- Simple Scale (Active Comparator): Individuals in this arm will receive standard care for their obesity in the Pediatric Weight Management Clinic and will be encouraged to self-weigh daily utilizing a simple scale.
  Interventions: Device: Simple Scale
- EHR-Connected Scale (Active Comparator): Individuals in this arm will receive standard care for their obesity in the Pediatric Weight Management Clinic and will be encouraged to self-weigh daily utilizing a Smart scale that is connected to the Electronic Health Record (EHR).
  Interventions: Device: EHR-Connected Scale

INTERVENTIONS:
Other: Standard Care — Individuals will receive standard care for their obesity through the Pediatric Weight Management Clinic.
  Arms: Standard Care
Device: Simple Scale — Individuals will be encouraged to perform daily weighing at home on a simple scale.
  Arms: Simple Scale
Device: EHR-Connected Scale — Individuals will be encouraged to perform daily weighing at home on a Smart scale that connects to the EHR. Clinic staff will review weight entries in the EHR and provide feedback.
  Arms: EHR-Connected Scale

SUMMARY:
99 patients age 12 to <18 years old with obesity (BMI >/=95th percentile), will be randomized to one of three treatment interventions:

1. Usual Care
2. Usual Care plus advice to weigh daily on simple scale
3. Usual Care plus advice to weigh-daily on an EHR-connected scale

Survey data collected at baseline, 2, 4, 6, and 12-weeks, and qualitative interviews at 12 weeks, will assess acceptability, safety, self-efficacy, and BMI. Recruitment will also be assessed (% eligible patients who consent). In order to understand real-world feasibility of this intervention, the clinic staff will work with patients to connect the scales to Epic.

DETAILED DESCRIPTION:
Obesity is a major public health issue because of its high prevalence and many health consequences. Obesity is driven by a dysregulation of the body's energy regulatory systems and is life-shortening. Obesity during the critical adolescent period increases risk of diabetes, cardiometabolic disease, all-cause mortality, and adulthood obesity. Rates of obesity-related cancers are increasing in younger populations. In addition to poorer health, individuals with obesity during adolescence are at risk for lower productivity, income, and likelihood of employment in adulthood, making obesity treatment and prevention important for reducing disparities. Despite consensus on the need for multi-component interventions for obesity, rates continue to climb for adolescents, youth of low-income backgrounds, and youth of racial/ethnic minority backgrounds. Clinicians cite lack of time and tools to help patients lose weight as barriers to weight counseling, and thus need practical, effective interventions they can feasibly disseminate from a busy clinical setting.

Self-weighing, grounded in behavior change theory, is effective for weight loss in adults. Self-monitoring is grounded in Social Cognitive Theory (SCT), which describes behavior change as happening with reciprocal interactions with one's environment, creating external and internal self-reinforcement. Self-monitoring is one such interaction that improves self-awareness through proximate self-measurement, and improves self-efficacy, self-control, and self-reinforcement. Self-weighing (SW) is a form of self-monitoring for weight loss that is grounded in SCT. Daily SW in adults has been associated with increased exercise and cognitive restraint, and reduced snacking, television watching, and consumption of sweets.

The investigator found no data on patient and parent perspectives on connecting scales to the EHR for daily weights in adolescents with obesity seeking obesity treatment.

99 patients age 12 to <18 years old with obesity (BMI >/=95th percentile), to be randomized to one of three treatment interventions:

1. Usual Care
2. Usual Care plus advice to weigh daily on simple scale
3. Usual Care plus advice to weigh-daily on an EHR-connected scale

Survey data collected at baseline, 2, 4, 6, and 12-weeks, and qualitative interviews at 12 weeks, will assess acceptability, safety, self-efficacy, and BMI. Recruitment will also be assessed (% eligible patients who consent). In order to understand real-world feasibility of this intervention, the clinic staff will work with patients to connect the scales to Epic.

ELIGIBILITY:
Inclusion Criteria for Adolescent:

* Ages 12 to < 18 years
* Body mass index (BMI) >/= 95th percentile

Exclusion Criteria for Adolescent:

* Score over 20 on the Eating Attitudes Test (EAT-26)
* Any unhealthy weight control behaviors
* Severe anxiety or depression
* Participation in another Pediatric Weight Management Clinic study
* Developmental delay
* Significant co-morbidity that might cause weight fluctuations in weight
* Current participation in a weight loss research study

Inclusion Criteria for Parent:

* Parent or legal guardian of the child participant
* Parent aged > 18 years

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 99 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of connecting the Smart scales to the EHR and access home weights through the EHR | 12 weeks
  Feasibility will be measured by determining if the clinic staff can successfully connect scales to the EHR and access home weights through the EHR. Staff will record time required to connect the scale, answer questions and trouble-shoot problems that arise with the scale between visits to understand the time burden of this intervention.
Feasibility of collecting daily weights. | 12 weeks
  Participants who are randomized to the simple scale and the EHR-connected scale will be asked to weigh themselves daily (which we anticipate will be 5-7 days per week). Participants who were randomized to the EHR-connected device will have their adherence measured by looking at the EHR to see how many daily weights were completed. Participants randomized to the simple scale will be self-reporting how many times per week they weighed themselves at home with the simple scale
Perceptions of daily weight tracking. | 12 weeks
  Participants who are randomized to perform daily weighing on a simple scale and on an EHR-connected scale will be asked about their perceptions of having to perform this task on a daily basis via a questionnaire. The questionnaire will be a Likert scale from 0 (not helpful, not motivated, not interesting, not satisfying) to 8 (extremely helpful, extremely motivated, extremely interesting, extremely satisfying).

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Bramante, MD, Principal Investigator — University of Minnesota
Locations (1):
- M Health - Pediatric Weight Management Clinic, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No